CLINICAL TRIAL: NCT02748083
Title: Research on Transcranial Direct Current Stimulation (tDCS) as a Treatment for Cognitive Deficits in Schizophrenic
Brief Title: Transcranial Direct Current Stimulation (tDCS) as a Treatment for Cognitive Deficits in Schizophrenic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Nathan Kline Institute for Psychiatric Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-09
Record Dates: First submitted 2016-01-15; First posted 2016-04-22 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Schizophrenia
Keywords: tDCS; schizophrenia; cognition; fMRI
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tDCS group (Active Comparator): The active tDCS group will be stimulated with transcranial Direct Current Stimulation (tDCS).
  Interventions: Device: tDCS
- Sham tDCS group (Sham Comparator): The sham tDCS group will have stimulation with sham transcranial Direct Current Stimulation (tDCS).
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: tDCS — Electrodes for tDCS will have the anode placed over the left DLPFC (F3) and the cathode over the contralateral (right) supraorbital ridge. The exact location of electrodes will be determined by the 10/20 EEG method with EEG cap. Subjects will have tDCS sessions on consecutive days (weekends and holidays excluded). The tDCS group will have 10 active or sham tDCS sessions. The active group will be stimulated with a 2 mA current for 20 minutes.
  Arms: tDCS group
Device: Sham tDCS — Electrodes for tDCS will have the anode placed over the left DLPFC (F3) and the cathode over the contralateral (right) supraorbital ridge. The exact location of electrodes will be determined by the 10/20 EEG method with EEG cap. Subjects will have tDCS sessions on consecutive days (weekends and holidays excluded). The sham tDCS group will have 10 active or sham tDCS sessions. The sham group will have stimulation lasting only 40 seconds though the electrodes will remain in place for 20 min.
  Arms: Sham tDCS group

SUMMARY:
This trial attempts to evaluate the effects of intensive transcranial direct-current stimulation (tDCS) on improving cognition in schizophrenia patients and changes in resting state brain network connectivity, especially increasing connectivity in the tasks related network, and increasing activation the DLPFC in a working memory task. Half of the participants will be randomized to tDCS group, while the other half will be randomized to receive sham tDCS.

DETAILED DESCRIPTION:
Schizophrenia patients (SZ) show profound and persistent cognitive deficits in attention, executive processing, and verbal and visuospatial memory, which persist even after psychotic symptoms are ameliorated. Cognitive deficits may be more important in preventing functional, occupational, and social recovery in SZ than other symptom domains and are not effectively treated by current pharmacological approaches. Transcranial direct-current stimulation (tDCS) is less expensive than other modalities (e.g. repetitive transcranial magnetic stimulation; rTMS), easily available, and has a good safety profile in healthy controls (HC) and SZ. However, these prior studies did not make use of a validated measure such as the MATRICS consensus battery (MCCB), which is now established as the standard for assessing cognitive improvement in SZ. Despite these promising preliminary results, this effect of tDCS in SZ needs to be confirmed and the underlying biological mechanism elucidated. Therefore, the investigators employed MCCB to evaluate the effects on improving cognition and functional MRI to explore the underlying mechanism.

Half of the participants will be randomized to tDCS group, while the other half will be randomized to receive sham tDCS. Active vs. sham treatment will be randomly using computer generated lists. Subjects and researcher-administrators of tDCS and testers or evaluators will be blind to treatment.The main cognitive outcome measure, the MCCB, will be administered at baseline and 1 day after the last tDCS session.Participants will be scanned once prior to tDCS sessions, and within one day after the 10th tDCS sessions using our Siemens 3T Verio MRI scanner.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have cognitive deficits as indicated by a score of < 85 on RBANS, and meet criteria for DSM-5 diagnosis of chronic SZ, schizoaffective disorder (SA), or schizophreniform disorder (SZF), and who are stably treated with antipsychotic medications and are not in acute exacerbation of illness symptoms.

Exclusion Criteria:

* Patients with risk factors for an MRI scan, seizure disorder, and for women of childbearing age who are pregnant or regularly engaging in sexual activity and not regularly using an acceptable birth control method (systemic or double-barrier).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
The MATRICS Consensus Cognitive Battery (MCCB) | Change from Baseline MCCB through study completion, an average of 15 days
Neuroimage changes in Magnetic Resonance Imaging (MRI) | Change from Baseline MCCB through study completion, an average of 15 days
  Including T1, resting state functional MRI, task based functional MRI and Diffusion Tensor Imaging(DTI)

SECONDARY OUTCOMES:
The CogState: Working memory and attention | through study completion, an average of 15 days
The Positive and Negative Syndrome Scale (PANSS) | Change from Baseline MCCB through study completion, an average of 15 days
Side-effects of tDCS | through study completion, an average of 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Chunbo Li, Ph.D., Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD data

REFERENCES:
- [Derived] Smith RC, Md WL, Wang Y, Jiang J, Wang J, Szabo V, Faull R, Jin H, Davis JM, Li C. Effects of transcranial direct current stimulation on cognition and symptoms in Chinese patients with schizophrenia✰. Psychiatry Res. 2020 Feb;284:112617. doi: 10.1016/j.psychres.2019.112617. Epub 2019 Nov 2. PMID 31806403